CLINICAL TRIAL: NCT05044494
Title: Surgery for Delay-recognized or Defer-operated Type A Aortic Dissection
Status: Completed | Type: Observational
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 21MMHIS005e
Record Dates: First submitted 2021-09-12; First posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-05

CONDITIONS: Aortic Dissection
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: non-prompt surgery after acute type a aortic dissection occurred
  Interventions: Procedure: non-prompt surgery
- control group: prompt surgery after acute type a aortic dissection occurred

INTERVENTIONS:
Procedure: non-prompt surgery
  Groups: study group

SUMMARY:
From November 2004 to June 2020, there were more than 200 patients with acute TAAD patients who underwent aortic surgery at our hospital.Of all the patients in the study period, there were 34 patients (defined as study group) who sought for medical attention with symptoms for several days (median 5 days, range 3-7 days) or deferred aortic surgery several days later (median 3 days, range 2-7 days) even though acute TAAD was diagnosed on the same day when chest pain or back pain occurred. For reducing the selection bias, propensity score matching (PSM) was used to match the study group with the control group from all the patients treated at our hospital during the study period. Comparison between the two groups was performed.

DETAILED DESCRIPTION:
From November 2004 to June 2020, there were more than 200 patients with acute TAAD patients who underwent aortic surgery at our hospital. The research protocol used in this study was approved by the institutional review board of MacKay Memorial Hospital (IRB number: 21MMHIS005e). Of all the patients in the study period, there were 34 patients (defined as study group) who sought for medical attention with symptoms for several days (median 5 days, range 3-7 days) or deferred aortic surgery several days later (median 3 days, range 2-7 days) even though acute TAAD was diagnosed on the same day when chest pain or back pain occurred. The mean age at presentation was 60.2 +/- 13.2 years (range 33.4~83.5 years). All the patients in the study group were divided into 3 groups: DP group (n=22) with acute TAAD diagnosis delayed by patient but received prompt aortic surgery; DD group (n=4) with acute TAAD diagnosis delayed by patient and received deferred aortic surgery; ID group (n=8) with acute TAAD diagnosis on the same day when the symptoms occurred but received deferred aortic surgery several days later. For reducing the selection bias, propensity score matching (PSM) was used to match the study group with the control group from all the patients treated at our hospital during the study period. Comparison between the two groups was performed.

ELIGIBILITY:
Inclusion Criteria:

* the patients sought for medical attention with symptoms (chest pain, back pain or shortness of breath) for several days or deferred aortic surgery several days later although acute TAAD was diagnosed on the same day when chest pain or back pain occurred

Exclusion Criteria:

-

Ages: 33 Years to 83 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: From November 2004 to June 2020, there were more than 200 consecutive patients with acute TAAD treated surgically at our hospital. Among all the acute TAAD patients, 34 patients sought for medical attention with symptoms (chest pain, back pain or shortness of breath) for several days or deferred aortic surgery several days later although acute TAAD was diagnosed on the same day when chest pain or back pain occurred.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2004-11; Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
surgical mortality | 2004-2020
  in-hospital death